CLINICAL TRIAL: NCT06575036
Title: Reversal of Rocuronium-induced Neuromuscular Blockade by Sugammadex in Children Younger Than 2 Years Old: a Prospective Dose Finding Study
Brief Title: Sugammadex Dose Finding Under Two Years Old
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sang-Hwan Ji (Other)
Responsible Party: Sponsor-Investigator, Sang-Hwan Ji, Clinical Assistant Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2308-161-1461
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Neuromuscular Blockade
Keywords: Sugammadex; Children; Dose-finding study
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: Up-and-down dose finding method using biased coin design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Sequential determination of dose according to previous participant's result and by chance.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — The starting dose of sugammadex will be 0.5mg/kg. When the dose for a patient was not effective, the dose for next patient will be increased by 0.5mg/kg. When the dose was effective, the dose for next patient will be decreased by 0.5mg/kg or maintained, with a 1:1 of allocation ratio.
  Other Names: Bridion

SUMMARY:
This is a prospective dose-finding study of sugammadex for conventional reversal of rocuronium-induced neuromuscular blockade in children under two years of age. This study will explore 50% effective dose and 95% effective dose of sugammadex for reversal of neuromuscular blockade in less than two minutes under biased coin up-and-down method.

DETAILED DESCRIPTION:
The investigators are planning to enroll 33 patients to obtain data. The starting dose of sugammadex will be 0.5mg/kg. When the dose for a patient was not effective, the dose for next patient will be increased by 0.5mg/kg. When the dose was effective, the dose for next patient will be decreased by 0.5mg/kg or maintained, with a 1:1 of allocation ratio.

The investigators will also monitor incidence of any adverse events including residual blockade to evaluate safety of sugammadex in children younger than two years old.

ELIGIBILITY:
Inclusion Criteria:

* Childern younger than 2 years old who are scheduled to undergo surgery under general anesthesia
* American Society of Anesthesiologists Physical Status 1 or 2

Exclusion Criteria:

* History of hypersensitivity to rocuronium or any anesthetics
* Presence of cardiovascular or genitourinary disease
* Presence of severe renal dysfunction or in need of dialysis
* Presence of severe hepatic dysfunction or coagualtion disorder
* Current state of administration of neuromuscular blocking agent on admission to operating room
* Concurrent use of any medications that affect the activity of neuromuscular blocking agents
* History of malignant hyperthermia
* Refusal to enroll in the study by one or more parents
* Presence of any other reasons that investigator regards inappropriate to enroll in the study.

Max Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
50% effective dose | From start of sugammadex administration to 2 minute after end of administration
  Dose of sugammadex that can reverse neuromuscular blockade in 50% of patients.
95% effective dose | From start of sugammadex administration to 2 minute after end of administration
  Dose of sugammadex that can reverse neuromuscular blockade in 95% of patients.

SECONDARY OUTCOMES:
TOF result | From start of sugammadex administration to 2 minute after end of administration
  Response to train-of-four stimulation after administration of sugammadex
Residual blockade | From start of sugammadex administration to 24 hours after end of administration
  Incidence of recurarization in the postanesthesia care unit
Blood pressure | From start of sugammadex administration to discharge from postanesthesia care unit (less than 3 hours)
  Noninvasive blood pressure after sugammadex administration measured in the operating room and postanesthesia care unit
Pulse oximetry | From start of sugammadex administration to discharge from postanesthesia care unit (less than 3 hours)
  Pulse oximetry after sugammadex administration measured in the operating room and postanesthesia care unit

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hwan Ji, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gijsenbergh F, Ramael S, Houwing N, van Iersel T. First human exposure of Org 25969, a novel agent to reverse the action of rocuronium bromide. Anesthesiology. 2005 Oct;103(4):695-703. doi: 10.1097/00000542-200510000-00007. PMID 16192761
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156
- [Background] Meibohm B, Laer S, Panetta JC, Barrett JS. Population pharmacokinetic studies in pediatrics: issues in design and analysis. AAPS J. 2005 Oct 5;7(2):E475-87. doi: 10.1208/aapsj070248. PMID 16353925
- [Background] Olutoye OA, Yu X, Govindan K, Tjia IM, East DL, Spearman R, Garcia PJ, Coulter-Nava C, Needham J, Abrams S, Kozinetz CA, Andropoulos DB, Watcha MF. The effect of obesity on the ED(95) of propofol for loss of consciousness in children and adolescents. Anesth Analg. 2012 Jul;115(1):147-53. doi: 10.1213/ANE.0b013e318256858f. Epub 2012 May 10. PMID 22575569
- [Background] Stylianou M, Flournoy N. Dose finding using the biased coin up-and-down design and isotonic regression. Biometrics. 2002 Mar;58(1):171-7. doi: 10.1111/j.0006-341x.2002.00171.x. PMID 11890313